CLINICAL TRIAL: NCT05664893
Title: Phase I/II Study to Determine the Safety and Efficacy of Ribociclib in Combination With Hormone Therapy and Hypofractionated Radiotherapy in Breast Cancer, With Positive Hormone Receptors and Negative HER2 Status, in Newly Diagnosed, Not Immediately Operable (or Wishing to Avoid Surgery), Elderly Patient (CALHYS)
Brief Title: Study to Determine the Safety and Efficacy of Ribociclib in Combination With Hormone Therapy and Hypofractionated Radiotherapy in Breast Cancer, With Positive Hormone Receptors and Negative HER2 Status, in Newly Diagnosed, Not Immediately Operable Elderly Patient (CALHYS)
Acronym: CALHYS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017/78
Record Dates: First submitted 2022-11-25; First posted 2022-12-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: HER2 Negative Breast Cancer Not Immediately Operated
MeSH Terms: interventions — ribociclib

STUDY DESIGN:
Intervention Model Description: step 1 : 600mg of ribociclib step 2 : 400mg of ribociclib step 3 : 200mg of ribociclib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Principal arm (Experimental): registration phase : 3 cycles of 600mg per day of ribociclib Treatment phase : 3 cycles of dose de-escalation of ribociclib (600 or 400 or 200mg per day) Maintenance phase : 600mg per day of ribociclib until 24months of total treatment
  Interventions: Drug: Ribociclib Oral Tablet

INTERVENTIONS:
Drug: Ribociclib Oral Tablet — 600mg per day during registration phase (3 cycles); de-escalation phase (600 to 200mg per day associated to radiotherapy) during 3 other cycles; maintenance phase until 24 months of treatment in total (600mg per day).
  All over th etimme, hormonotherapy is received in concomitance

SUMMARY:
Women aged 70 years or older, newly diagnosed for locally advanced unilateral breast cancer, with a histological diagnosis of invasive mammary carcinoma, positive hormone receptors, HER2 status Negative, not immediately operable (stage of disease, comorbidities or refusal of surgery) with tumor in place, with indication of treatment with hormone therapy and hypofractionated radiotherapy, not eligible for neoadjuvant chemotherapy and without major comorbidity contraindicating the proposed treatment regimen.

ELIGIBILITY:
Criteria for registration phase Inclusion criteria

1. Written informed consent must be obtained prior to any screening procedures;
2. Women ≥ 70 years old at the time of signing informed consent;
3. Have a performance status of 0 to 2 on the ECOG Performance Scale ;
4. Newly diagnosed for non-metastatic unilateral breast cancer;
5. Histological diagnosis of invasive mammary carcinoma, positive hormone receptors, HER2 status Negative defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing and based on the most recently analyzed tissue sample;
6. Not immediately operable (stage of disease, comorbidities or wish to avoid surgery) with tumor in place;
7. Measurable disease based on RECIST 1.1 (a lesion at a previously irradiated site may only be counted as a target lesion if there is a clear sign of progression since the irradiation).
8. Demonstrate adequate organ functions:

   1. Hemoglobin > 9 g/dL;
   2. Absolute neutrophil count > 1.5 G/L;
   3. Platelets > 100 G/L;
   4. INR ≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug);
   5. Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN in patients with well documented Gilbert's Syndrome
   6. AST and ALT < 2.5 x ULN;
   7. Alkaline Phosphatase < 2.5 x ULN
   8. Calculated creatinine clearance > 30 ml/min using MDRD formula;
   9. Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements (the local laboratory value should be documented within normal limits after the correction) before registration:

      * Potassium
      * Magnesium
      * Total Calcium (corrected for serum albumin);
9. Standard 12-lead ECG values defined as the mean of the triplicate ECGs

   * QTcF interval at screening < 450 msec (QT interval using Fridericia's correction)
   * Mean resting heart rate 50-90 bpm (determined from the ECG)
10. Indication of treatment with hormone therapy and hypofractioned radiotherapy;
11. Patients having taken cognizance of the information sheet and having signed the informed consent;
12. Patients covered by medical insurance.
13. Must be able to swallow ribociclib;
14. Subjects must be able to communicate with the investigator and comply with the requirements of the study procedures;
15. Must be willing to remain at the clinical site as required by the protocol.

Exclusion criteria

1. Patient eligible to resection surgery and wish to proceed with the surgery;
2. Patient eligible to neoadjuvant chemotherapy;
3. Patient with distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition);
4. Concomitant bilateral breast cancer;
5. Previous treatment, in the 2 years before inclusion, by chemotherapy, hormone therapy (more than 6 months before study registration), thoracic surgery or radiotherapy for a malignant tumor;
6. Tumor in previously irradiated territory;
7. Patient has received any CDK4/6 inhibitor;
8. Patient with a known hypersensitivity to any of the excipients of Ribociclib and/or hormono therapy (e.g. rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, glucose-galactose malabsorption, and soy allergy);
9. Known additional malignancy. Exceptions include basal cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy;
10. Contraindication for hormone therapy , Ribociclib or radiotherapy;
11. Severe dementia;
12. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
13. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol: (e.g., chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)

    * Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:
    * History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
    * Documented cardiomyopathy
    * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
    * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug)
    * Inability to determine the QTcF interval
    * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
    * Systolic Blood Pressure (SBP) >160 or <90 mmHg
14. Patient is currently receiving any of the following substances within 7 days before randomization:

    1. Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pomelos, starfruit, Seville oranges) and their juices that are known as strong inhibitors or inducers of CYP3A4/5;
    2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5;
15. Vulnerable persons as defined by article L1121-5 - 8:

    1. Pregnant women, women in labor or breast-feeding mothers, persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8
    2. Persons admitted to a social or health facility for reasons other than research;
    3. Adults subject to a legal protection order or unable to give their consent.
16. Concurrent enrolment in another clinical trial using an investigational anti-cancer treatment within 28 days prior to the first dose of study treatment.

Criteria for the Ribociclib and Radiotherapy concomitant phase Inclusion criteria

1. Patient registered in the study-screening phase;
2. Patient receiving, during the registration phase, 3 cycles of Ribociclib at 600mg without dose decreased;
3. Have a performance status of 0 to 2 on the ECOG Performance Scale;
4. Not immediately operable (stage of disease, comorbidities or refusal of surgery) with tumor in place;
5. Measurable disease based on RECIST 1.1;
6. Demonstrate adequate organ functions:

   1. Hemoglobin > 9 g/dL;
   2. Absolute neutrophil count > 1.5 G/L;
   3. Platelets > 100 G/L;
   4. INR ≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug);
   5. Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN; in patients with well documented Gilbert's Syndrome;
   6. AST and ALT <2.5 x ULN;
   7. Alkaline Phosphatase < 2.5 x ULN
   8. Calculated creatinine clearance > 30 ml/min using MDRD formula;
   9. Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements (the local laboratory value should be documented within normal limits after the correction) before inclusion:

      * Potassium
      * Magnesium
      * Total Calcium (corrected for serum albumin);
7. Standard 12-lead ECG values defined as the mean of the triplicate ECGs

   * QTcF interval at screening < 450 msec (QT interval using Fridericia's correction)
   * Mean resting heart rate 50-90 bpm (determined from the ECG)Indication of treatment with hormone therapy and hypofractioned radiotherapy;
8. Patients having taken cognizance of the information sheet and having signed the informed consent;
9. Patients covered by medical insurance.
10. Must be able to swallow ribociclib;
11. Subjects must be able to communicate with the investigator and comply with the requirements of the study procedures;
12. Must be willing to remain at the clinical site as required by the protocol.

Exclusion criteria

1. Patient eligible to resection surgery after 3 cycles of Ribociclib;
2. Patient eligible to neoadjuvant chemotherapy;
3. Concomitant bilateral breast cancer;
4. Known additional malignancy. Exceptions include basal cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy;
5. Contraindication for hormone therapy, Ribobociblib or radiotherapy;
6. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol: (e.g., chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)

   * Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:
   * History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
   * Documented cardiomyopathy
   * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
   * Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
   * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug)
   * Inability to determine the QTcF interval
   * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
   * Systolic Blood Pressure (SBP) >160 or <90 mmHg
7. Severe dementia;
8. Patients unable to express their consent;
9. Vulnerable persons as defined by article L1121-5 - 8:

   1. Pregnant women, women in labor or breast-feeding mothers, persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8;
   2. Persons admitted to a social or health facility for reasons other than research;
   3. Adults subject to a legal protection order or unable to give their consent.
10. Concurrent enrolment in another clinical trial using an investigational anti-cancer treatment.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Phase I : determination of Maximal Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D) of Ribociclib | Phase I : during the 8 weeks of radiotherapy concomitant with the Ribociclib and hormone therapy and during the 3 months of post-radiotherapy follow-up.
  Phase I : the frequencies of adverse events according to the CTCAE 4.03 requiring a dose discontinuation (DLT) will be determined during the 8 weeks of radiotherapy concomitant with the Ribociclib and hormone therapy and during the 3 months of post-radiotherapy follow-up.
Phase II : evaluation of the efficacy of Ribociclib in association with hormone therapy and hypofractionated radiotherapy | Phase II : at 24-months
  Phase II :The primary endpoint will be the rate of non-progression at 24-months, defined as the percentage of patients who are alive and have not progressed 24 months after the completion of the Ribociclib and Radiotherapy concomitant phase.

SECONDARY OUTCOMES:
overall survival | 24 months
  Evaluate overall survival (OS)
overall survival | 60 months
  Evaluate overall survival (OS)
progression free survival | 24 months
  Evaluate progression free survival (PFS)
progression free survival | 60 months
  Evaluate progression free survival (PFS)
quality of Life (European Organisation for Research and Treatment of Cancer quality of life questionnaire C30) | 60 months
  Evaluate quality of Life (items values from 1 to 4 per question)
quality of Life (ELDERLY CANCER PATIENTS14) | 60 months
  Evaluate quality of Life (items values from 1 to 4 per question)
compliance to Ribociclib | 24 months
  The treatment compliance will be assessed with the 8-item Morisky Medication Adherence Scale (score from 0 to 8)
medical health status | 60 months
  Evaluate the medical health status of the patients with the questionnaire G8, clinical score and visual analog scale for pain severity measurement (score from 0 to 17)
psychosocial health status | 60 months
  Evaluate the psychosocial status of the patients with GDS 4 questionnaire (score from 0 to 4)
functional health status | 60 months
  Evaluate the functional status of the patients with the questionnaires MINI MENTAL STATE EXAMINATION (score from 0 to 30)
functional health status | 60 months
  Evaluate the functional status of the patients with the questionnaires Autonomy Daily Living (score from 0 to 6)
functional health status | 60 months
  Evaluate the functional status of the patients with the questionnaires (Instrumental Activities in Daily Living (score from 0 to 8)
functional health status | 60 months
  Evaluate the functional status of the patients with the questionnaires walking speed
functional health status | 60 months
  Evaluate the functional status of the patients with the questionnaires percentage of weight loss
functional health status | 60 months
  Evaluate the functional status of the patients with Handgrip strength evaluation
overall tolerance of ribociclib using V5.0 Common Terminology Criteria for Adverse Events scale | 25 months
  The overall tolerance of Ribociclib during ribociclib monotherapy treatment and concomitant ribociclib radiotherapy treatment will be evaluated using clinical and biological assessment and graded according to the V5.0 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No